CLINICAL TRIAL: NCT03757949
Title: A Randomized Phase III Double Blind Clinical Trial Evaluating the Effect of Immune-Enhancing Nutrition on Radical Cystectomy Outcomes
Brief Title: Nutrition Therapy in Improving Immune System in Patients With Bladder Cancer That Can Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: S1600; NCI-2017-02442 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1600 (Other: SWOG); SWOG-S1600 (Other: DCP); S1600 (Other: CTEP); UG1CA189974 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-11-29 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (SIM) (Experimental): Patients receive SIM PO TID on days -5 to -1 and 1-5. Patients undergo standard of care surgery on day 0.
  Interventions: Other: Laboratory Biomarker Analysis; Dietary Supplement: Nutritional Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): ARM II: Patients receive placebo PO TID on days -5 to -1 and 1-5. Patients undergo standard of care surgery on day 0.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Dietary Supplement: Nutritional Intervention — Receive SIM PO
  Arms: Arm I (SIM)
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well nutrition therapy works in improving immune system in patients with bladder cancer that can be removed by surgery. Improving nutrition before and after surgery may reduce the infections and other problems that sometimes occur after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the impact of consuming perioperative specialized immune-modulating drinks (SIM, Impact Advanced Recovery, Nestle) to oral nutrition supplement control drinks (ONS, Oral Nutrition Control, Nestle) on post-operative complications (any versus [vs.] none) within 30 days after scheduled radical cystectomy (RC).

SECONDARY OBJECTIVES:

I. To assess whether SIM use compared to ONS reduces late-phase post-operative complications within 90 days after scheduled RC.

II. To assess whether SIM use compared to ONS reduces infections. III. To assess whether SIM use compared to ONS reduces skeletal muscle wasting. IV. To assess whether SIM use compared to ONS reduces high grade post-operative complications.

V. To assess whether SIM use compared to ONS reduces readmission rates. VI. To assess whether SIM use compared to ONS improves quality of life. VII. To assess whether SIM use compared to ONS improves disease-free survival after surgery and overall survival.

TERTIARY OBJECTIVES:

I. To assess the impact of SIM use on the expansion of myeloid-derived suppressor cells.

II. To assess the impact of SIM use on pro-inflammatory cytokines and neutrophil: lymphocyte ratios.

III. To assess the impact of SIM use on post-operative arginine deficiency and amino acid metabolism.

IV. To explore the association of dietary intake variables (nutrition status, calories, protein, and immune-enhancing factors) and study outcomes.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To describe the microbiome of the gut in patients undergoing radical cystectomy and urinary diversion prior to initiation of immunonutrition or a nutrition control.

II. To define the microbiome change in patients undergoing radical cystectomy and urinary diversion after they have received blinded immunonutrition or control nutritional supplement.

III. To correlate cancer treatments, postoperative complications (specifically infections) and nutritional status with microbiome composition.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive SIM orally (PO) thrice daily (TID) on days -5 to -1 and 1-5. Patients undergo standard of care surgery on day 0.

ARM II: Patients receive placebo PO TID on days -5 to -1 and 1-5. Patients undergo standard of care surgery on day 0.

After completion of study, patients are followed up at 2, 30, and 90 days, and at 6, 9, 12, 18, 24, and 36 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a tissue diagnosis of primary cell carcinoma of the bladder by transurethral resection of bladder tumor (TURBT) or partial cystectomy; patients may not have any evidence of unresectable disease or metastatic disease as assessed by exam under anesthesia or imaging (computed tomography [CT], magnetic resonance imaging [MRI], positron-emission tomography [PET])
* There must be plans for the cystectomy to be performed within 28 calendar days after registration
* Surgery must be planned to be performed under pre-approved, study-specific surgical guidelines
* Patients must have completed any neoadjuvant chemotherapy or immunotherapy (intravesical or systemic) >= 14 calendar days prior to registration and any toxicities resolved to at least grade 2
* Patients may have a history of radiation therapy; radiation therapy must have been completed >= 180 days prior to registration
* Patients may have a history of prior partial cystectomy; prior partial cystectomy must have been completed at least 180 days prior to registration
* Patients with planned adjuvant chemotherapy within 90 days after radical cystectomy will not be eligible
* Patients must be able to swallow liquid and have no refractory nausea, vomiting, malabsorption, or significant small bowel resection that would preclude adequate absorption; patients on tube feeding are not eligible
* Patients must have their baseline nutrition status assessed using the Scored Patient-Generated Subjective Global Assessment (PG-SGA) by a clinician or licensed healthcare practitioner (trained physician, nurse, or dietician) within 14 days prior to registration and must not have a global category rating of stage C (severely malnourished)
* Patients must not have galactosemia
* Patients must not have known active viral infections such as human immunodeficiency virus (HIV) or hepatitis, as these chronic viral infections may cause cachexia and immunodeficiency and thus alter the biology regarding the study endpoints
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for two years; prostate cancer found at cystectomy would not be considered a prior malignancy
* Patients must not be pregnant or nursing as the conditions preclude candidacy for radical cystectomy
* Patients must consent and be willing to have specimens collected and submitted
* Patients must be offered the opportunity to participate in additional specimen banking
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients must consent and provide their telephone contact information for four 24-hour dietary recall phone interviews to be conducted by staff at the Exercise, Diet, Genitourinary, & Endocrinology Laboratory (EDGE) Research Laboratory
* Patients must be able to understand and speak English and/or Spanish because the dietary recall phone interviews will only be conducted in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2027-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Hamilton-Reeves, Principal Investigator — SWOG Cancer Research Network
Locations (46):
- United States (46):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Rochester, Rochester, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (SIM) | Arm II (Placebo)
Started | 99 | 104
Completed | 90 | 88
Not Completed | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (SIM) | Arm II (Placebo) | Total
Number analyzed (Participants) | 99 | 104 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 66 | 72 | 138
Age, Continuous [Median (Full Range); unit: years] | 68 [41.4 to 90.6] | 69.45 [32 to 95.2] | 68.8 [32 to 95.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 77 | 85 | 162
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 6 | 10
  White | 68 | 79 | 147
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 17 | 39
Region of Enrollment [Number; unit: participants]
  United States | 99 | 104 | 203

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Complications
Description: A post-operative complication is defined as a binary indicator variable indicating whether the patient experienced any complication (any/none; Clavien-Dindo grades I-V). The primary analysis will be based on a multivariable logistic regression under intent-totreat among all randomized patients, irrespective of their eligibility status, adjusting for the specified stratification factors: a. Diversion type (neobladder versus [vs.] ileal conduit); b. Prior neoadjuvant chemotherapy (any vs. none); and c. Nutrition status (well nourished vs. moderate malnutrition). A Fisher's exact test will also be conducted to establish whether the results are sensitive to model assumptions. A single interim analysis for efficacy will be conducted when 50% of patients achieve their endpoint at the alpha=0.005 level. Accordingly, the final analysis will be conducted at the alpha=0.045 level. A separate analysis among all eligible randomized patients will also be conducted.
Time Frame: Up to 30 days post surgery
Population: Participants who are evaluable at day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (SIM) | Arm II (Placebo)
Number analyzed (Participants) | 90 | 88
Participants | 56 | 51

2. Secondary Outcome: Post-Op Complications
Time Frame: This outcome measure will be reported by 9/28/2025
Reporting Status: Not Posted, anticipated posting 2025-09

3. Secondary Outcome: Infections
Time Frame: This outcome measure will be reported by 9/28/2025
Reporting Status: Not Posted, anticipated posting 2025-09

4. Secondary Outcome: Skeletal Muscle Wasting
Time Frame: This outcome measure will be reported by 9/28/2025
Reporting Status: Not Posted, anticipated posting 2025-09

5. Secondary Outcome: High Grade Post-Op Complications
Time Frame: This outcome measure will be reported by 9/28/2025
Reporting Status: Not Posted, anticipated posting 2025-09

6. Secondary Outcome: Readmission Rates
Time Frame: This outcome measure will be reported by 9/28/2025
Reporting Status: Not Posted, anticipated posting 2025-09

7. Secondary Outcome: Quality of Life
Time Frame: This outcome measure will be reported by 9/28/2025
Reporting Status: Not Posted, anticipated posting 2025-09

8. Secondary Outcome: Disease Free Survival
Time Frame: This outcome measure will be reported by 9/28/2025
Reporting Status: Not Posted, anticipated posting 2025-09

ADVERSE EVENTS:
Time Frame: Once within 14 days after preoperative treatment, once within 14 days after post-operative treatment.
Description: Adverse Events are assessed using CTCAE version 5.0.
  The population assessed is not the same as analysis population. The analysis population was among all randomized (not just eligible participants), with evaluability based on assessment for primary outcome. Whereas the AE/SAE population was all eligible patients, assessed for AEs, and evaluable for survival endpoints.
Groups:
- Arm I (SIM): Patients receive SIM PO TID on days -5 to -1 and 1-5. Patients undergo standard of care surgery on day 0.XXXLaboratory Biomarker Analysis: Correlative studiesXXXNutritional Intervention: Receive SIM POXXXQuality-of-Life Assessment: Ancillary studiesXXXQuestionnaire Administration: Ancillary studies
- Arm II (Placebo): ARM II: Patients receive placebo PO TID on days -5 to -1 and 1-5. Patients undergo standard of care surgery on day 0.XXXLaboratory Biomarker Analysis: Correlative studiesXXXPlacebo Administration: Given POXXXQuality-of-Life Assessment: Ancillary studiesXXXQuestionnaire Administration: Ancillary studies
Arm/Group | Arm I (SIM) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 9/91 | 17/88
Serious Adverse Events (participants affected / at risk) | 2/91 | 2/88
Other Adverse Events (participants affected / at risk) | 68/91 | 67/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (SIM) (N=91) | Arm II (Placebo) (N=88)
Cardiac arrest (Cardiac disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (SIM) (N=91) | Arm II (Placebo) (N=88)
Anemia (Blood and lymphatic system disorders) | 18 | 21
Leukocytosis (Blood and lymphatic system disorders) | 6 | 5
Sinus tachycardia (Cardiac disorders) | 5 | 4
Abdominal distension (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 16 | 17
Bloating (Gastrointestinal disorders) | 8 | 7
Constipation (Gastrointestinal disorders) | 15 | 12
Diarrhea (Gastrointestinal disorders) | 17 | 9
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 4 | 7
Ileus (Gastrointestinal disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 28 | 26
Vomiting (Gastrointestinal disorders) | 20 | 14
Chills (General disorders) | 6 | 2
Edema limbs (General disorders) | 5 | 7
Fatigue (General disorders) | 14 | 16
Fever (General disorders) | 15 | 4
Pain (General disorders) | 15 | 7
Sepsis (Infections and infestations) | 5 | 3
Urinary tract infection (Infections and infestations) | 19 | 10
Creatinine increased (Investigations) | 10 | 11
Anorexia (Metabolism and nutrition disorders) | 6 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 6
Hypokalemia (Metabolism and nutrition disorders) | 6 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 8 | 5
Hyponatremia (Metabolism and nutrition disorders) | 8 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 4
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Dizziness (Nervous system disorders) | 7 | 3
Hematuria (Renal and urinary disorders) | 6 | 4
Renal and urinary disorders-Other (Renal and urinary disorders) | 6 | 4
Hypertension (Vascular disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT03757949/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT03757949/ICF_001.pdf